CLINICAL TRIAL: NCT04127864
Title: Perioperative Immune Function in Patients Undergoing Colorectal Cancer Surgery Using a Functional Whole Blood Immune Stimulation Assay
Brief Title: Perioperative Immune Function in Patients Undergoing Colorectal Cancer Surgery
Acronym: TruCulture
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Rune Børch Hasselager, Principal Investigator, Zealand University Hospital
Other Study IDs: TruCulture
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal cancer surgery — All participants will undergo surgery for colorectal cancer.

SUMMARY:
At Zealand University Hospital, Denmark, the investigators will examine the immune function of patients with colorectal cancer before and after tumor resection.

The immune function will be assessed with functional profiling of the immune function (TruCulture®)

The study aims to describe alterations in the perioperative immune response to surgery. The generatied knowledge will lead to better under standing of perioperative pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic resection of colorectal cancer with curative intent

Exclusion Criteria:

* Age under 18
* Neoadjuvant chemo or radiation therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for minimally invasive colorectal cancer resection at Zealand University Hospital. They will undergo standard treatment characterized by strict adherence to the enhanced recovery after surgery guidelines
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Cytokines in LPS stimulated blood | Postoperative day 1
  Difference in cytokine levels (interleukin-1b(IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-7 (IL-7), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-12 70p (IL-12 (70)), interleukin-13 (IL-13), interleukin-17 (IL-17), Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) interpheron-gamme (IFN-γ), monocyte chemoattractant protein 1 (MCP-1), Macrophage inflammatory protein-1β (MIP-1β), tumor necrosis factor alpha (TNF-α) all pg/ml) between postoperative and preoperative whole blood exposed to lipopolysaccharide measured with multiplex assay (Bio-Plex Pro™ Human Cytokine 17-plex Assay (M50-00031YV) by Bio-Rad)
Cytokines in CD3+CD28 stimulated blood | Postoperative day 1
  Difference in cytokine levels (interleukin-1b(IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-7 (IL-7), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-12 70p (IL-12 (70)), interleukin-13 (IL-13), interleukin-17 (IL-17), Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) interpheron-gamme (IFN-γ), monocyte chemoattractant protein 1 (MCP-1), Macrophage inflammatory protein-1β (MIP-1β), tumor necrosis factor alpha (TNF-α) all pg/ml) between postoperative and preoperative whole blood exposed to CD3 and CD28 measured with multiplex assay (Bio-Plex Pro™ Human Cytokine 17-plex Assay (M50-00031YV) by Bio-Rad)
Cytokines in Poly I:P stimulated blood | Postoperative day 1
  Difference in cytokine levels (interleukin-1b(IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-7 (IL-7), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-12 70p (IL-12 (70)), interleukin-13 (IL-13), interleukin-17 (IL-17), Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) interpheron-gamme (IFN-γ), monocyte chemoattractant protein 1 (MCP-1), Macrophage inflammatory protein-1β (MIP-1β), tumor necrosis factor alpha (TNF-α) all pg/ml) between postoperative and preoperative whole blood exposed to Polyinosinic:polycytidylic acid measured with multiplex assay (Bio-Plex Pro™ Human Cytokine 17-plex Assay (M50-00031YV) by Bio-Rad)
Cytokines in R848 stimulated blood | Postoperative day 1
  Difference in cytokine levels (interleukin-1b(IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-7 (IL-7), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-12 70p (IL-12 (70)), interleukin-13 (IL-13), interleukin-17 (IL-17), Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) interpheron-gamme (IFN-γ), monocyte chemoattractant protein 1 (MCP-1), Macrophage inflammatory protein-1β (MIP-1β), tumor necrosis factor alpha (TNF-α) all pg/ml) between postoperative and preoperative whole blood exposed to Resiquimod (R848) measured with multiplex assay (Bio-Plex Pro™ Human Cytokine 17-plex Assay (M50-00031YV) by Bio-Rad)

SECONDARY OUTCOMES:
Cytokines in unstimulated blood | Postoperative day 1
  Difference in cytokine levels (interleukin-1b(IL-1β), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5), interleukin-6 (IL-6), interleukin-7 (IL-7), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-12 70p (IL-12 (70)), interleukin-13 (IL-13), interleukin-17 (IL-17), Granulocyte colony-stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF) interpheron-gamme (IFN-γ), monocyte chemoattractant protein 1 (MCP-1), Macrophage inflammatory protein-1β (MIP-1β), tumor necrosis factor alpha (TNF-α) all pg/ml) between postoperative and preoperative plasma measured with multiplex assay (Bio-Plex Pro™ Human Cytokine 17-plex Assay (M50-00031YV) by Bio-Rad)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, DMSc, Study Director — Center for Surgical Science, Zealand University Hospital, Denmark
Locations (1):
- Center for Surgical Science, Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided